CLINICAL TRIAL: NCT07391644
Title: A First-in-Human, Open-Label, Multicenter, Phase 1 Study to Evaluate the Safety, Tolerability, and Preliminary Antitumor Activity of JSKN027 in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of JSKN027 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSKN027-101
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JSKN027 (Experimental): Participants will receive JSKN027 administered by intravenous infusion at dose levels based on actual body weight (mg/kg). The planned dose levels are 1, 3, 6, 10, 15, and 20 mg/kg, administered once every 3 weeks (Q3W).
  Interventions: Drug: JSKN027

INTERVENTIONS:
Drug: JSKN027 — JSKN027 is an investigational therapeutic agent being evaluated for the treatment of advanced malignant solid tumors. It is administered as intravenous monotherapy at multiple dose levels in this study.

SUMMARY:
This is a first-in-human, open-label, multicenter Phase 1 (Ia/Ib) clinical study conducted in China to evaluate the safety and tolerability of JSKN027 in patients with advanced malignant solid tumors. The study will also assess the pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of JSKN027, and determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D).

The study includes two parts. Part Ia is a dose-escalation phase designed to evaluate the safety and tolerability of increasing dose levels of JSKN027. Part Ib is a dose-expansion phase in which additional patients will be enrolled at selected dose levels to further evaluate safety and preliminary antitumor activity in specific tumor types. Initial expansion cohorts are planned for patients with colorectal cancer, non-small cell lung cancer, and hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, multicenter Phase 1 (Ia/Ib) clinical study conducted in China to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of JSKN027 in patients with advanced malignant solid tumors, and to determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D).

The study consists of two parts: a dose-escalation phase (Part Ia) and a dose-expansion phase (Part Ib). In Part Ia, an accelerated titration design followed by an i3+3 dose-escalation design will be used to evaluate multiple dose levels of JSKN027 and assess its safety and tolerability. In Part Ib, multiple expansion cohorts will be enrolled based on tumor type to further evaluate the safety and preliminary efficacy of JSKN027 at selected dose levels. Initial expansion cohorts are planned for patients with colorectal cancer (CRC), non-small cell lung cancer (NSCLC), and hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of signing the ICF.
* ECOG performance status 0-1.
* Estimated life expectancy ≥ 3 months.
* Histologically or cytologically confirmed advanced or metastatic malignant solid tumor.
* For dose escalation (Part Ia): disease has progressed on standard therapy.
* For dose expansion (Part Ib): participants with prespecified tumor types (e.g., colorectal cancer, non-small cell lung cancer, hepatocellular carcinoma, and other selected solid tumors) who have progressed on standard therapy.
* At least one measurable extracranial lesion per RECIST v1.1.
* Adequate bone marrow function within 7 days prior to enrollment (e.g., ANC ≥ 1.5×10^9/L, hemoglobin ≥ 90 g/L, platelets ≥ 100×10^9/L).
* Adequate hepatic function within 7 days prior to enrollment (e.g., total bilirubin, AST/ALT, ALP within protocol-defined limits; albumin ≥ 30 g/L).
* Adequate renal function within 7 days prior to enrollment (e.g., serum creatinine ≤ 1.5×ULN or creatinine clearance ≥ 60 mL/min; urine protein within acceptable limits).
* Adequate coagulation function within 7 days prior to enrollment (e.g., PT/INR and aPTT within protocol-defined limits).
* Adequate cardiac function (e.g., LVEF ≥ 50%).
* Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.
* Participants of reproductive potential agree to use highly effective contraception from ICF signing until 7 months after the last dose.

Exclusion Criteria:

* Active central nervous system (CNS) disease (e.g., active brain metastases or leptomeningeal disease).
* Received an investigational agent within 28 days or 5 half-lives (whichever is shorter) prior to first dose.
* Major surgery within 28 days prior to first dose or planned major surgery during the study.
* History of severe immune-related adverse events or prior toxicity that would preclude safe participation, as judged by the investigator.
* Significant gastrointestinal disorders that increase risk of perforation, bleeding, obstruction, or interfere with study participation.
* Active or uncontrolled interstitial lung disease (ILD) or non-infectious pneumonitis, or suspected ILD/pneumonitis at screening.
* Active autoimmune disease requiring systemic immunosuppression (exceptions may apply for limited, stable conditions).
* Active hepatitis B or C, HIV infection, or other clinically significant immunodeficiency/infection not adequately controlled per local standards.
* Prior allogeneic organ or bone marrow transplant.
* Known hypersensitivity to the study drug or its excipients, or history of severe hypersensitivity to similar biologic agents.
* Pregnant or breastfeeding.
* Any condition that, in the investigator's judgment, would compromise participant safety or compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose-Limiting Toxicities (DLTs) | From first dose of JSKN027 through 21 days after the first dose (DLT evaluation period)
  The number of participants who experience dose-limiting toxicities (DLTs) during the dose-limiting toxicity evaluation period following administration of JSKN027
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From first dose of JSKN027 through 30 days after the last dose
  The number of participants who experience treatment-emergent adverse events (TEAEs) following administration of JSKN027, graded according to NCI CTCAE version 5.0.
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of JSKN027 | From first dose of JSKN027 through completion of dose-escalation phase (approximately 12 months)
  Determination of the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of JSKN027 based on observed dose-limiting toxicities and overall safety and tolerability.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by RECIST v1.1 | From first dose of JSKN027 until disease progression or death, up to 24 months
  Objective response rate (ORR), defined as the proportion of participants with a best overall response of complete response (CR) or partial response (PR), as assessed by the investigator according to RECIST version 1.1.
Disease Control Rate (DCR) as Assessed by RECIST v1.1 | From first dose of JSKN027 until disease progression or death, up to 24 months
  Disease control rate (DCR), defined as the proportion of participants with a best overall response of complete response (CR), partial response (PR), or stable disease (SD), as assessed by the investigator according to RECIST version 1.1.
Duration of Response (DoR) as Assessed by RECIST v1.1 | From first documented response until disease progression or death, up to 24 months
  Duration of response (DoR), defined as the time from first documented objective response (CR or PR) to disease progression or death, as assessed according to RECIST version 1.1.
Progression-Free Survival (PFS) | From first dose of JSKN027 until disease progression or death, up to 24 months
  Progression-free survival (PFS), defined as the time from first dose of JSKN027 to the first documentation of disease progression or death from any cause.
Overall Survival (OS) | From first dose of JSKN027 until death from any cause, up to 36 months
  Overall survival (OS), defined as the time from first dose of JSKN027 to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No